CLINICAL TRIAL: NCT03779074
Title: Efficacies of Hybrid, High-dose Dual and Bismuth Quadruple Therapies for the First-line Anti-H Pylori Treatment and Tetracycline-levofloxacin Quadruple Therapy for the Second-line Anti-H Pylori Treatment - a Multicentre Randomized Trial
Brief Title: Comparing the Efficacy of Hybrid, High-dose Dual and Bismuth Quadruple Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS18-CT4-24
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication rate
MeSH Terms: interventions — Rabeprazole; BID protein, human; Tetracycline; Metronidazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10d bismuth quadruple therapy (Active Comparator): rabeprazole 20 mg b.i.d. plus tripotassium dicitrate bismuthate 300 mg, tetracycline 500 mg and metronidazole 250 mg q.i.d. for 10 days.
  Interventions: Drug: 10d bismuth quadruple therapy
- 14d hybrid therapy (Experimental): a dual regimen with rabeprazole 20 mg and amoxicillin 1 g b.i.d. for 7 days followed by a quadruple regimen with rabeprazole 20 mg, amoxicillin 1 g, clarithromycin 500 mg and metronidazole 500 mg b.i.d. for 7 days.
  Interventions: Drug: 14d hybrid therapy
- 14d high-dose dual therapy (Experimental): rabeprazole 20 mg and amoxicillin 750 mg q.i.d. for 14 days
  Interventions: Drug: 14D high-dose dual therapy

INTERVENTIONS:
Drug: 10d bismuth quadruple therapy — rabeprazole 20 mg b.i.d. plus tripotassium dicitrate bismuthate 300 mg, tetracycline 500 mg and metronidazole 250 mg q.i.d. for 10 days
  Other Names: rabeprazole 20 mg bid; tripotassium dicitrate bismuthate 300mg qid; tetracycline 500 mg qid; metronidazole 250 mg qid
  Arms: 10d bismuth quadruple therapy
Drug: 14d hybrid therapy — a dual regimen with rabeprazole 20 mg and amoxicillin 1 g b.i.d. for 7 days followed by a quadruple regimen with rabeprazole 20 mg, amoxicillin 1 g, clarithromycin 500 mg and metronidazole 500 mg b.i.d. for 7 days
  Other Names: rabeprazole 20 mg bid; amoxicillin 1 g bid; clarithromycin 500 mg bid; metronidazole 500 mg bid
  Arms: 14d hybrid therapy
Drug: 14D high-dose dual therapy — rabeprazole 20 mg and amoxicillin 750 mg q.i.d. for 14 days
  Other Names: rabeprazole 20 mg qid; amoxicillin 750 mg qid
  Arms: 14d high-dose dual therapy

SUMMARY:
Both hybrid and high-dose dual therapies developed by the scholars from Taiwan can achieve a high eradication rate for clarithromycin-resistant strains, and have a great potential to replace bismuth quadruple therapy in the treatment of H. pylori infection.

DETAILED DESCRIPTION:
Bismuth quadruple therapy has been recommended as a choice of the first-line treatment for H. pylori infection in several important international consensuses. However, it is associated with a high frequency of adverse events. Both hybrid and high-dose dual therapies developed by the scholars from Taiwan can achieve a high eradication rate for clarithromycin-resistant strains, and have a great potential to replace bismuth quadruple therapy in the treatment of H. pylori infection. In the second-line treatment, tetracycline-levofloxacin quadruple therapy developed by our study group can achieve a higher eradication rate than levofloxacin triple therapy for salvage treatment of hybrid therapy. However, whether the new therapy can be a promising rescue treatment for bismuth quadruple or high-dose dual therapy remains unanswered.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H pylori-infected outpatients, at least 20 years of age, with endoscopically proven peptic ulcer diseases or gastritis

Exclusion Criteria:

* previous H pylori-eradication therapy
* ingestion of antibiotics or bismuth within the prior 4 weeks
* patients with allergic history to the medications used
* patients with previous gastric surgery
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 918 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants in Which H. Pylori Was Eradicated | sixth week after the end of anti- H. pylori therapy
  To assess eradication efficacy with urea breath test

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu PI, Chen KY, Tai WC, Yang JC, Tsay FW, Liu YH, Chen CL, Lee CL, Yeh HZ, Kuo CH, Chuah SK, Lee HC, Shie CB, Shiu SI, Kao JY, Yamaoka Y, Graham DY, Wu DC; Taiwan Acid-related Disease (TARD) Study Group. Hybrid, High-Dose Dual and Bismuth Quadruple Therapies for First-Line Treatment of Helicobacter pylori Infection in Taiwan: A Multicenter, Open-Label, Randomized Trial. Am J Gastroenterol. 2023 Jul 1;118(7):1184-1195. doi: 10.14309/ajg.0000000000002255. Epub 2023 Mar 20. PMID 36940437